CLINICAL TRIAL: NCT01620892
Title: Outcomes of Patients With Unicompartmental Arthritis of the Knee Five Years After Treatment With Partial Knee Replacement
Brief Title: Study of Patient Outcomes 5 Years After Partial Knee Replacement
Status: Completed | Type: Observational
Sponsor: Athens Orthopedic Clinic, P.A. (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Ormonde M. Mahoney, MD, Principal Investigator, Orthopedic Surgeon, Athens Orthopedic Clinic, P.A.
Other Study IDs: AOC-OM-Arthrex-001
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: unicondylar knee arthroplasty; partial knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unicondylar knee replacement: This is a non-intervational, retrospective, observational study of a case series cohort of patients who received a particular surgical operation during a specified time period.

SUMMARY:
The study seeks to evaluate the condition of patients 5 years after having undergone partial knee replacement for localized osteoarthritis of the knee. Participating patients will voluntarily undergo detailed evaluation of clinical and radiologic outcomes 5 years after surgery. The aims of the study are to describe the survivorship of the prostheses and the clinical results of patients, and to elucidate and describe the natural history disease of the untreated knee joint compartments after a partial replacement. Patients who were operated by the principal investigator 5 years previously will be invited to participate. The study is observational in nature; there is no element of experimentation or test of an intervention.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who have undergone unicondylar knee replacement of a single tibio-femoral compartment using iBalance prosthesis (Arthrex, Inc, Lakeland Florida) under the care of the principal investigator between December, 2006 and December, 2008 will be invited to participate in the study.

Exclusion Criteria:

* There are no restrictions to inclusion in the study based on surgical or medical criteria; however, individuals who are pregnant, incarcerated, less than 18 years of age, or unable to give valid informed consent on their own behalf will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential study population consists of all patients who have undergone implantation of a specific unicondylar knee arthroplasty device under the care of the principal investigator between December, 2006 and December, 2008. This is a clinic-based sample of consecutive cases.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to revision of the partial total knee prosthesis | 5 to 7 years after original implantation
  Eligible participants are invited to enroll into this observational study after the 5-year anniversary of the index primary knee replacement procedure. The participant will be evaluated once to determine whether the original implant is in situ, or has been revised. Method of determination will include self-report of the participant, medical records review/verification, and radiographic examination of the prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Ormonde M Mahoney, MD, Principal Investigator — Athens Orthopedic Clinic, P.A.
Locations (1):
- Athens Orthopedic Clinic, P.A., Athens, Georgia, United States